CLINICAL TRIAL: NCT07032935
Title: The Effect of Virtual Reality Glasses on Vital Signs and State Anxiety in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KutahyaHSU20240106
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Coronary Angiography (CAG)
Keywords: coronary angiography; virtual reality glasses; anxiety; vital signs
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: virtual reality glasses
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention will be made to the patient during the Coronary Angiography application.
- virtual reality glasses Group (Experimental)
  Interventions: Behavioral: Virtual Reality Glasses will be used DURING CORONARY ANGIOGRAPHY APPLICATION

INTERVENTIONS:
Behavioral: Virtual Reality Glasses will be used DURING CORONARY ANGIOGRAPHY APPLICATION — Virtual Reality Glasses will be used DURING CORONARY ANGIOGRAPHY APPLICATION
  Arms: virtual reality glasses Group

SUMMARY:
Virtual reality (VR) glasses are an effective non-pharmacological method for reducing anxiety, supported by a high level of evidence and associated with no known side effects. Techniques involving relaxation and distraction, such as VR, function by suppressing the sympathetic branch of the autonomic nervous system and activating the parasympathetic branch, thereby eliciting a relaxation response.

VR glasses divert the patient's attention away from pain and anxiety. By reducing the sense of unfamiliarity in clinical environments, VR helps patients adapt more easily, leading to enhanced relaxation. This state of relaxation not only alleviates anxiety but also induces favorable physiological responses. These include reductions in blood pressure (BP), heart rate (HR), and respiratory rate (RR), along with an increase in peripheral oxygen saturation (SpO₂). Additionally, the psychological benefits of VR contribute to the reduction of anxiety, stress, fear, and worry.

VR is considered a cost-effective, safe, and non-pharmacological intervention. Several studies support its efficacy. For example, in a study comparing the effects of video games played through VR headsets and iPads on preoperative anxiety in adult patients undergoing sternotomy, anxiety was measured using the Depression Anxiety Stress Scale (DASS), and lower anxiety levels were observed in the VR group. Another study demonstrated that watching nature scenes through VR glasses for five minutes prior to maxillofacial surgery significantly reduced anxiety. Furthermore, research comparing progressive muscle relaxation exercises and VR during arthroscopic knee surgery-measured using the State Anxiety Inventory-indicated that both non-pharmacological interventions were effective in reducing anxiety.

However, despite this growing body of evidence, no study to date has examined the effects of VR applications on anxiety in patients undergoing coronary angiography or pacemaker implantation. This study aims to fill that gap by investigating the comparative effectiveness of virtual reality applications in reducing anxiety in patients undergoing coronary angiography.

ELIGIBILITY:
Inclusion Criteria: Patients who will undergo coronary angiography or pacemaker implantation, Not to receive sedation during the procedure, Written and verbal acceptance to participate in the study,

* Are over 18 years of age,
* Do not have any psychiatric illness,
* Do not have any vision, hearing or perception problems,
* Are at least a primary school graduate,
* Do not have any disorder/disease affecting decision-making ability (dementia, psychological disorder, etc.)
* Volunteer to participate in the study,
* Are open to communication and cooperation.

Exclusion Criteria:

* Patients who receive sedation, patients who cannot communicate, patients with visual or hearing impairments, and individuals who do not agree to participate in the research will be included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Score | Before the intervention (15 minutes before the procedure), and within the first 15 minutes after the intervention is completed
  Before and after the intervention (pre- and post-intervention) It will be measured using the State Anxiety Inventory (STAI-I). The score varies between 20 and 80.

SECONDARY OUTCOMES:
Change in Vital Signs (Heart Rate) | Before the intervention (15 minutes before the procedure), and within the first 15 minutes after the intervention is completed
  To be measured before and after the virtual reality intervention
Change in Vital Signs (Blood Pressure) | Before the intervention (15 minutes before the procedure), and within the first 15 minutes after the intervention is completed
  To be measured before and after the virtual reality intervention
Change in Vital Signs (Respiratory Rate) | Before the intervention (15 minutes before the procedure), and within the first 15 minutes after the intervention is completed
  To be measured before and after the virtual reality intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No